CLINICAL TRIAL: NCT05148793
Title: A Clinical Examination of N95 Reuse and Extended Use
Brief Title: N95 Reuse During COVID-19
Acronym: ReuseN95
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, San Diego (Other); Johns Hopkins University (Other); University of Wisconsin, Madison (Other); Emory University (Other); University of Rochester (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 21-33232
Record Dates: First submitted 2021-12-06; First posted 2021-12-08 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Emergency Medicine; Frontline Providers; Healthcare Worker
Keywords: N95 mask; Personal Protective Equipment; Extended use; reuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During critical personal protective equipment (PPE) shortages, such as those associated with the COVID-19 pandemic, Centers for Disease Control (CDC) recommends N95 extended use (wearing the same N95 for multiple patient encounters) and limited reuse (storing an N95 between shifts for use over multiple shifts with or without decontamination) as contingency and crisis capacity strategies, respectively. Many healthcare workers (HCWs) are employing these strategies out of necessity. The sustained performance of these respirators depends on the respirator maintaining its filtration efficiency and its ability to provide an adequate seal (fit) to the user's face. Fit testing is performed when a respirator is issued to the user and on an annual basis thereafter. A user-seal check is then performed whenever a respirator is donned. Previous studies have found repeated donnings/doffings to significantly decrease the respirator's fit. A recent pilot cross-sectional clinical study conducted by the University of California, San Francisco found fit failures of respirators after being worn for 2 shifts. However, more definitive data regarding respirator performance during reuse and extended use are lacking. The investigators plan to address these critical gaps in knowledge by conducting a prospective cohort study to determine the incidence of N95 fit failure when subjected to extended use/reuse in a clinical setting. The investigators plan to enroll 396 ED providers (including physicians, nurses, and staff) when obtaining a new NIOSH approved N95s and performing serial fit tests at the end of each 8-12 hour shift for up to 5 clinical shifts or until N95 failure, whichever is earlier. By carefully measuring fit test failure in a clinical setting, the investigators will be able to provide guidance regarding the safety of N95 extended use and reuse necessitated by the need for PPE conservation. Specifically, the investigators will address the following research questions: 1) how long N95s maintain their fit during extended use, 2) how many times N95s can be donned/doffed and maintain their fit, 3) the ability of a user seal check to indicate fit in the field, 4) what adverse health effects, reports of discomfort, or symptoms are experienced by users during extended use and reuse, 5) what effect does extended use and reuse have on N95 filtration performance, 6) the level of contamination of N95s when subjected to extended use and reuse, 7) the effect of modifications to N95 (covering an N95 with a face shield or surgical N95s, facial coverings) on fit failure.

DETAILED DESCRIPTION:
Frontline healthcare workers are at high risk of SARS (severe acute respiratory syndrome) CoV-2 (COVID-19) infection. Personal protective equipment (PPE), such as an N95 respirator (N95), is essential for prevention of COVID-19 among HCWs. N95s can prevent aerosolized transmission of viral particles and reduce COVID-19 among HCWs, helping to reduce infection rates and preserve the workforce. Under normal circumstances, the CDC recommends that HCWs dispose of N95s after a single patient encounter. However, during critical PPE shortages such as those during the current COVID-19 pandemic, the CDC recommends N95 extended use (wearing the same N95 for multiple patient encounters) and re-use (storing an N95 between shifts for use over multiple shifts). N95 shortages have been widely reported during the COVID-19 pandemic and have forced HCWs to practice extended use and reuse of N95s. Despite the CDC's guidelines, there are limited data regarding the efficacy of N95s under conditions of extended use and reuse and existing studies have been conducted in laboratory settings rather than in the actual health care environment. (Bergman 2012; Vuma et al 2019). This has left health care workers, including emergency department (ED) providers on the front lines of the COVID-19 pandemic, without clear guidance regarding N95 conservation. Many have implemented various reuse and extended use policies out of necessity but with no empirical evidence of their safety and effectiveness.

The study team conducted a pilot cross-sectional study of 68 ED providers who wore either a 3M 1860 dome style N95 or a duckbill N951. 70.6% of duckbill N95 failed a standardized fit test with 3M bitter solution and a hood. Of the dome style , 27.5% failed a fit test. N95 failure was associated with increasing numbers of shifts used: There were 0/11 failures after 1 shift, 1/12 failures after 2 shifts, 3/13 failures after 3 shifts, and 10/15 failures after 4 or more shifts. Also, more donnings and doffings were associated with fit failure, with a median of 8 donning and doffings in the fit pass group and 15 donning and doffings in the fit failure group. This preliminary study had a number of limitations, including a small sample size, convenience sampling, and cross-sectional design, and so was unable to definitively identify the number of shifts or donnings/doffings for which N95s can be safely reused.

The investigators propose to conduct a prospective cohort study of 396 participants across 6 ED sites to estimate the cumulative incidence of N95s when subjected to extended use and reuse in a clinical (emergency department) setting with fit test failure and contamination as the main endpoints. The investigators also seek to compare the fit test failure between varying types of HCWs wearing a number of N95 types. Additionally, the investigators will collect the N95s used in this study for additional analyses of at an outside laboratory measuring COVID-19 contamination levels and filtration efficiency.

ELIGIBILITY:
Inclusion criteria

* Adult (18 years old or greater)
* ED providers (MDs, nurses, Advanced Practice Providers (APPs)) who are practicing extended use and re-use for the majority (more than half) of their shifts Participants are eligible when obtaining a new N95 and are scheduled to work a minimum of 5 shifts within a 60-day period. As hours of enrollment and data collection depend on research associate availability, participants working certain shifts may not be eligible.

Exclusion criteria:

* Participant does not intend to use N95 for majority of shift
* Schedule prohibits re-use and or data collection
* Repeated failed baseline fit test
* Refused or unable to consent
* Pregnant
* Facial hair (e.g., beards or sideburns) or jewelry which interferes with the face seal region of an N95

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare provider, specifically frontline workers that involves direct patient contact.
Sampling Method: Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with qualitative fit test failure (N95 A, end of shift 1) | At the end of shift A1, up to 12 hours
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 1, for N95 A. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).
Number of participants with qualitative fit test failure (N95 A, end of shift 2) | At the end of shift A2, up to 12 hours per shift, 24 hours maximum
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 2, for N95 A. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).
Number of participants with qualitative fit test failure (N95 A, end of shift 3) | At the end of shift A3, up to 12 hours per shift, 36 hours maximum
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 3, for N95 A. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).
Number of participants with qualitative fit test failure (N95 A, end of shift 4) | At the end of shift A4, up to 12 hours per shift, 48 hours maximum
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 4, for N95 A. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).
Number of participants with qualitative fit test failure (N95 A, end of shift 5) | At the end of shift A5, up to 12 hours per shift, 60 hours maximum
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 5, for N95 A. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).
Number of participants with qualitative fit test failure (N95 B, end of shift 1) | At the end of shift B1, up to 12 hours maximum
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 1, for N95 B. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).
Number of participants with qualitative fit test failure (N95 B, end of shift 2) | At the end of shift B2, up to 12 hours per shift, 24 hours maximum
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 2, for N95 B. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).
Number of participants with qualitative fit test failure (N95 B, end of shift 3) | At the end of shift B3, up to 12 hours per shift, 36 hours maximum
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 3, for N95 B. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).
Number of participants with qualitative fit test failure (N95 B, end of shift 4) | At the end of shift B4, up to 12 hours per shift, 48 hours maximum
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 4, for N95 B. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).
Number of participants with qualitative fit test failure (N95 B, end of shift 5) | At the end of shift B5, up to 12 hours per shift, 60 hours maximum
  Qualitative fit test outcome is measured by a trained fit tester at the end of participant shift 5, for N95 B. The fit test is performed up to 5 times per N95 or until fit test failure. The fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no).

SECONDARY OUTCOMES:
Number of participants with User Seal Check failure (N95 A, end of shift 1) | At the end of shift A1, up to 12 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given facial filtering respirator (FFR) develops an acceptable "leak-free" seal with a subject's face. A user seal check (USC) is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research Clinical Research Coordinator (CRC) will record whether the user seal check indicates a good seal.
Number of participants with User Seal Check failure (N95 A, end of shift 2) | At the end of shift A2, up to 12 hours per shift, 24 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given FFR develops an acceptable "leak-free" seal with a subject's face. A USC is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research CRC will record whether the user seal check indicates a good seal.
Number of participants with User Seal Check failure (N95 A, end of shift 3) | At the end of shift A3, up to 12 hours per shift, 36 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given FFR develops an acceptable "leak-free" seal with a subject's face. A USC is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research CRC will record whether the user seal check indicates a good seal.
Number of participants with User Seal Check failure (N95 A, end of shift 4) | At the end of shift A4, up to 12 hours per shift, 48 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given FFR develops an acceptable "leak-free" seal with a subject's face. A USC is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research CRC will record whether the user seal check indicates a good seal.
Number of participants with User Seal Check failure (N95 A, end of shift 5) | At the end of shift A5, up to 12 hours per shift, 60 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given FFR develops an acceptable "leak-free" seal with a subject's face. A USC is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research CRC will record whether the user seal check indicates a good seal.
Number of participants with User Seal Check failure (N95 B, end of shift 1) | At the end of shift B1, up to 12 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given FFR develops an acceptable "leak-free" seal with a subject's face. A USC is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research CRC will record whether the user seal check indicates a good seal.
Number of participants with User Seal Check failure (N95 B, end of shift 2) | At the end of shift B2, up to 12 hours per shift, 24 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given FFR develops an acceptable "leak-free" seal with a subject's face. A USC is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research CRC will record whether the user seal check indicates a good seal.
Number of participants with User Seal Check failure (N95 B, end of shift 3) | At the end of shift B3, up to 12 hours per shift, 36 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given FFR develops an acceptable "leak-free" seal with a subject's face. A USC is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research CRC will record whether the user seal check indicates a good seal.
Number of participants with User Seal Check failure (N95 B, end of shift 4) | At the end of shift B4, up to 12 hours per shift, 48 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given FFR develops an acceptable "leak-free" seal with a subject's face. A USC is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research CRC will record whether the user seal check indicates a good seal.
Number of participants with User Seal Check failure (N95 B, end of shift 5) | At the end of shift B5, up to 12 hours per shift, 60 hours maximum
  Participants will be asked to perform a brief "self- test" occurring prior to an actual fit test to determine that a given FFR develops an acceptable "leak-free" seal with a subject's face. A USC is subjective and determines whether the participant feels that the respirator seals well enough with the participant's face to proceed forward with the actual fit test. The research CRC will record whether the user seal check indicates a good seal.

OTHER OUTCOMES:
Number of participants with qualitative fit test failure of Mask A (at Baseline) | Prior to study inclusion
  Qualitative fit test outcome for Mask A is measured by a trained fit tester prior to study inclusion. For each of the 2 N95s, the fit tester records whether the N95 passed fit testing (Yes or No). The fit test variable outcome indicates a passed fit test (yes) or failed fit test (no). Only passed N95s may continue into the study. Failed mask details (manufacturer, lot number, expiration date) are collected for analysis.
N95 B Outcome | Within 6 months of enrollment
  N95 Qualitative Fit Test Outcome is measured over a maximum of 5 study shifts per N95. An Study N95s B can have 1 of 3 outcomes: (1) Passed all 5 fit tests, (2) Failed before 5 fit tests, or (3) Experienced Competing Event. N95s that either pass all 5 fit tests or experience a competing event which precludes the N95 from being fit tested will be censored in Kaplan Meier curve analysis.
N95 A Outcome | Within 6 months of enrollment
  N95 Qualitative Fit Test Outcome is measured over a maximum of 5 study shifts per N95. A Study N95s A can have 1 of 3 outcomes: (1) Passed all 5 fit tests, (2) Failed before 5 fit tests, or (3) Experienced Competing Event. N95s that either pass all 5 fit tests or experience a competing event which precludes the N95 from being fit tested will be censored in Kaplan Meier curve analysis.
N95 contamination as measured by Real-time Quantitative Polymerase Chain Reaction (RTqPCR) for COVID-19 (to be assessed by collecting masks and sending out to lab) | At the end of all study shifts, up to 10 visits (60 hours maximum).
  Each N95 labeled 'Mask A' which fails or is censored (completes 5 shifts or experiences competing event) will be collected in a sealable plastic storage container, stored, and shipped to Applied Research Associates.
N95 filtration as measured using TSI 8130, measuring flow rate (ml/min), particle penetration (%), and pressure drop (mmH2O). | At the end of all study shifts, up to 10 visits (60 hours maximum).
  Each N95 labeled 'Mask B' which fails or is censored (completes 5 shifts or experiences competing event) will be collected in a sealable plastic storage container, stored, and shipped to Applied Research Associates.
Participant reported symptoms (comfort) | At the end of each shift, up to 12 hours
  The investigators will collect data on participant reported outcomes, including symptoms from survey of participants at end of each shift, using the validated R-COMFI scale to measure mask discomfort.
Number of N95 donnings and doffings for Mask A during shift 1 (N95 A, end of shift 1) | At the end of shift A1, up to 12 hours maximum
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of N95 donnings and doffings for Mask A during shift 2 (N95 A, end of shift 2) | At the end of shift A2, up to 12 hours per shift, 24 hours maximum
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of N95 donnings and doffings for Mask A during shift 3 (N95 A, end of shift 3) | At the end of shift A3, up to 12 hours per shift, 36 hours maximum
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of N95 donnings and doffings for Mask A during shift 4 (N95 A, end of shift 4) | At the end of shift A4, up to 12 hours per shift, 48 hours maximum
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of N95 donnings and doffings for Mask A during shift 5 (N95 A, end of shift 5) | At the end of shift A5, up to 12 hours per shift, 60 hours maximum
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of N95 donnings and doffings for Mask B during shift 1 (N95 B, end of shift 1) | At the end of shift B1, up to 12 hours
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of N95 donnings and doffings for Mask B during shift 2 (N95 B, end of shift 2) | At the end of shift B2, up to 12 hours
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of N95 donnings and doffings for Mask B during shift 3 (N95 B, end of shift 3) | At the end of shift B3, up to 12 hours
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of N95 donnings and doffings for Mask B during shift 4 (N95 B, end of shift 4) | At the end of shift B4, up to 12 hours
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of N95 donnings and doffings for Mask B during shift 5 (N95 B, end of shift 5) | At the end of shift B5, up to 12 hours
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of total N95 donnings and doffings for Mask A during shifts 1-5 | Cumulative donning/doffing for up to 5 shifts, up to 12 hours each shift.
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Number of total N95 donnings and doffings for Mask B during shifts 1-5 | Cumulative donning/doffing for up to 5 shifts, up to 12 hours each shift.
  When a mask is removed and replaced on the face to be worn, participants will count 1 "donning & doffing".
Shift Length (N95 A, end of shift 1) | At the end of shift A1, up to 12 hours per shift.
  Length of participant's shift in hours.
Shift Length (N95 A, end of shift 2) | At the end of shift A2, up to 12 hours per shift.
  Length of participant's shift in hours.
Shift Length (N95 A, end of shift 3) | At the end of shift A3, up to 12 hours per shift.
  Length of participant's shift in hours.
Shift Length (N95 A, end of shift 4) | At the end of shift A4, up to 12 hours per shift.
  Length of participant's shift in hours.
Shift Length (N95 A, end of shift 5) | At the end of shift A5, up to 12 hours per shift.
  Length of participant's shift in hours.
Shift Length (N95 B, end of shift 1) | At the end of shift B1, up to 12 hours per shift.
  Length of participant's shift in hours.
Shift Length (N95 B, end of shift 2) | At the end of shift B2, up to 12 hours per shift.
  Length of participant's shift in hours.
Shift Length (N95 B, end of shift 3) | At the end of shift B3, up to 12 hours per shift.
  Length of participant's shift in hours.
Shift Length (N95 B, end of shift 4) | At the end of shift B4, up to 12 hours per shift.
  Length of participant's shift in hours.
Shift Length (N95 B, end of shift 5) | At the end of shift B5, up to 12 hours per shift.
  Length of participant's shift in hours.
Cumulative Shift Length (N95 A) | Up to 5 shifts, up to 12 hours per shift.
  Total length of participant's shifts in hours.
Cumulative Shift Length (N95 B) | Up to 5 shifts, up to 12 hours per shift.
  Total length of participant's shifts in hours.
Estimated Hours Worn (N95 A, end of shift 1) | At the end of shift A1, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Estimated Hours Worn (N95 A, end of shift 2) | At the end of shift A2, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Estimated Hours Worn (N95 A, end of shift 3) | At the end of shift A3, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Estimated Hours Worn (N95 A, end of shift 4) | At the end of shift A4, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Estimated Hours Worn (N95 A, end of shift 5) | At the end of shift A5, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Estimated Hours Worn (N95 B, end of shift 1) | At the end of shift B1, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Estimated Hours Worn (N95 B, end of shift 2) | At the end of shift B2, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Estimated Hours Worn (N95 B, end of shift 3) | At the end of shift B3, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Estimated Hours Worn (N95 B, end of shift 4) | At the end of shift B4, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Estimated Hours Worn (N95 B, end of shift 5) | At the end of shift B5, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Cumulative Estimated Hours Worn (N95 A) | Total estimated hours worn for up to 5 shifts, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Cumulative Estimated Hours Worn (N95 B) | Total estimated hours worn for up to 5 shifts, up to 12 hours per shift.
  Participants will estimate the total hours the N95 was worn.
Tightness of Straps, A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Tightness of Straps, A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Tightness of Straps, A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Tightness of Straps, A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Tightness of Straps, A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Tightness of Straps, B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Tightness of Straps, B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Tightness of Straps, B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Tightness of Straps, B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Tightness of Straps, B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to tightness of straps during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Irritation, B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial irritation (leaves marks/indents) during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Itching, B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial itching during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Pinching, B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial pinching during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nose, nose-bridge (pinching, redness from metal band), B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nose and nose-bridge pinching/redness from metal band during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Facial Heat/Warmth, B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to facial heat/warmth during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Sweat/Moisture buildup, B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to sweat/moisture buildup during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Lack of Fresh Air, B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to lack of fresh air during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Nausea, B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to nausea during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, A1 | At the end of shift A1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, A2 | At the end of shift A2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, A3 | At the end of shift A3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, A4 | At the end of shift A4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, A5 | At the end of shift A5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, B1 | At the end of shift B1, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, B2 | At the end of shift B2, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, B3 | At the end of shift B3, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, B4 | At the end of shift B4, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Headache, B5 | At the end of shift B5, up to 12 hours
  Level of N95 discomfort as measured by how often wearing the fit-tested filtering face-piece respirator caused discomfort due to headache during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, A1 | At the end of shift A1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, A2 | At the end of shift A2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, A3 | At the end of shift A3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, A4 | At the end of shift A4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, A5 | At the end of shift A5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, B1 | At the end of shift B1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, B2 | At the end of shift B2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, B3 | At the end of shift B3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, B4 | At the end of shift B4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dizziness, B5 | At the end of shift B5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dizziness during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, A1 | At the end of shift A1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, A2 | At the end of shift A2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, A3 | At the end of shift A3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, A4 | At the end of shift A4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, A5 | At the end of shift A5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, B1 | At the end of shift B1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, B2 | At the end of shift B2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, B3 | At the end of shift B3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, B4 | At the end of shift B4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Loss of energy/tiredness/fatigue, B5 | At the end of shift B5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting loss of energy/tiredness/fatigue during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, A1 | At the end of shift A1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, A2 | At the end of shift A2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, A3 | At the end of shift A3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, A4 | At the end of shift A4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, A5 | At the end of shift A5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, B1 | At the end of shift B1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, B2 | At the end of shift B2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, B3 | At the end of shift B3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, B4 | At the end of shift B4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Claustrophobia, B5 | At the end of shift B5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting claustrophobia during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, A1 | At the end of shift A1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, A2 | At the end of shift A2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, A3 | At the end of shift A3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, A4 | At the end of shift A4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, A5 | At the end of shift A5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, B1 | At the end of shift B1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, B2 | At the end of shift B2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, B3 | At the end of shift B3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, B4 | At the end of shift B4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Shortness of Breath, B5 | At the end of shift B5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting shortness of breath during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, A1 | At the end of shift A1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, A2 | At the end of shift A2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, A3 | At the end of shift A3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, A4 | At the end of shift A4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, A5 | At the end of shift A5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, B1 | At the end of shift B1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, B2 | At the end of shift B2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, B3 | At the end of shift B3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, B4 | At the end of shift B4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Difficulty Breathing, B5 | At the end of shift B5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting difficulty breathing during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, A1 | At the end of shift A1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift A1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, A2 | At the end of shift A2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift A2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, A3 | At the end of shift A3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift A3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, A4 | At the end of shift A4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift A4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, A5 | At the end of shift A5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift A5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, B1 | At the end of shift B1, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift B1. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, B2 | At the end of shift B2, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift B2. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, B3 | At the end of shift B3, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift B3. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, B4 | At the end of shift B4, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift B4. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Dry or Itchy Eyes, B5 | At the end of shift B5, up to 12 hours
  Qualitative experience of wearing N95 as measured by participant reporting dry or itchy eyes during shift B5. R-COMFI scaled variable with three potential outcomes, in order of increasing severity: none of the time, some of the time, all of the time.
Concentration, A1 | At the end of shift A1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift A1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Concentration, A2 | At the end of shift A2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift A2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Concentration, A3 | At the end of shift A3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift A3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Concentration, A4 | At the end of shift A4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift A4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Concentration, A5 | At the end of shift A5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift A5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Concentration, B1 | At the end of shift B1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift B1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Concentration, B2 | At the end of shift B2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift B2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Concentration, B3 | At the end of shift B3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift B3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Concentration, B4 | At the end of shift B4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift B4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Concentration, B5 | At the end of shift B5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask affected my concentration while working (always adjusting the mask)" during shift B5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, A1 | At the end of shift A1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift A1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, A2 | At the end of shift A2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift A2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, A3 | At the end of shift A3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift A3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, A4 | At the end of shift A4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift A4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, A5 | At the end of shift A5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift A5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, B1 | At the end of shift B1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift B1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, B2 | At the end of shift B2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift B2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, B3 | At the end of shift B3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift B3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, B4 | At the end of shift B4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift B4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Verbally Communicate, B5 | At the end of shift B5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficulty verbally communicating to others (unintelligible, muffled speech)" during shift B5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, A1 | At the end of shift A1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift A1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, A2 | At the end of shift A2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift A2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, A3 | At the end of shift A3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift A3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, A4 | At the end of shift A4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift A4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, A5 | At the end of shift A5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift A5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, B1 | At the end of shift B1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift B1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, B2 | At the end of shift B2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift B2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, B3 | At the end of shift B3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift B3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, B4 | At the end of shift B4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift B4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Hearing, B5 | At the end of shift B5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "I had difficultly hearing others" during shift B5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, A1 | At the end of shift A1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift A1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, A2 | At the end of shift A2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift A2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, A3 | At the end of shift A3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift A3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, A4 | At the end of shift A4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift A4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, A5 | At the end of shift A5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift A5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, B1 | At the end of shift B1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift B1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, B2 | At the end of shift B2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift B2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, B3 | At the end of shift B3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift B3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, B4 | At the end of shift B4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift B4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Obstructed Vision, B5 | At the end of shift B5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask obstructed my vision" during shift B5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, A1 | At the end of shift A1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift A1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, A2 | At the end of shift A2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift A2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, A3 | At the end of shift A3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift A3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, A4 | At the end of shift A4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift A4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, A5 | At the end of shift A5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift A5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, B1 | At the end of shift B1, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift B1. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, B2 | At the end of shift B2, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift B2. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, B3 | At the end of shift B3, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift B3. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, B4 | At the end of shift B4, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift B4. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Interfered Care, B5 | At the end of shift B5, up to 12 hours
  Qualitative assessment of N95 functionality as measured by participant reporting their level of agreement with the statement "The mask interfered with my patient care duties (quick to leave room, less interaction)" during shift B5. R-COMFI scaled variable with four potential outcomes, in order of increasing severity: strongly disagree, disagree, agree, strongly agree.
Irritated Skin, A1 | At the end of shift A1, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift A1.
Irritated Skin, A2 | At the end of shift A2, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift A2.
Irritated Skin, A3 | At the end of shift A3, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift A3.
Irritated Skin, A4 | At the end of shift A4, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift A4.
Irritated Skin, A5 | At the end of shift A5, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift A5.
Irritated Skin, B1 | At the end of shift B1, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift B1.
Irritated Skin, B2 | At the end of shift B2, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift B2.
Irritated Skin, B3 | At the end of shift B3, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift B3.
Irritated Skin, B4 | At the end of shift B4, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift B4.
Irritated Skin, B5 | At the end of shift B5, up to 12 hours
  Assessment of any facial irritation/marks/dents as measured by photographic evidence after shift B5.
Facial Thermal Sensation, A1 | At the end of shift A1, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift A1 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Facial Thermal Sensation, A2 | At the end of shift A2, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift A2 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Facial Thermal Sensation, A3 | At the end of shift A3, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift A3 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Facial Thermal Sensation, A4 | At the end of shift A4, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift A4 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Facial Thermal Sensation, A5 | At the end of shift A5, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift A5 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Facial Thermal Sensation, B1 | At the end of shift B1, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift B1 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Facial Thermal Sensation, B2 | At the end of shift B2, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift B2 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Facial Thermal Sensation, B3 | At the end of shift B3, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift B3 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Facial Thermal Sensation, B4 | At the end of shift B4, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift B4 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Facial Thermal Sensation, B5 | At the end of shift B5, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their face during shift B5 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, A1 | At the end of shift A1, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift A1 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, A2 | At the end of shift A2, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift A2 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, A3 | At the end of shift A3, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift A3 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, A4 | At the end of shift A4, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift A4 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, A5 | At the end of shift A5, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift A5 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, B1 | At the end of shift B1, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift B1 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, B2 | At the end of shift B2, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift B2 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, B3 | At the end of shift B3, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift B3 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, B4 | At the end of shift B4, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift B4 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Body Thermal Sensation, B5 | At the end of shift B5, up to 12 hours
  Qualitative assessment of N95 comfort measured by participant reporting of the thermal sensation of their whole body during shift B5 as very hot, hot, warm, slightly warm, neither warm nor cool, slightly cool, cool, cold, very cold.
Aerosolized Generating Procedures, A1 | At the end of shift A1, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, cardiopulmonary resuscitation (CPR), respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift A1.
Aerosolized Generating Procedures, A2 | At the end of shift A2, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, CPR, respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift A2.
Aerosolized Generating Procedures, A3 | At the end of shift A3, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, CPR, respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift A3.
Aerosolized Generating Procedures, A4 | At the end of shift A4, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, CPR, respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift A4.
Aerosolized Generating Procedures, A5 | At the end of shift A5, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, CPR, respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift A5.
Aerosolized Generating Procedures, B1 | At the end of shift B1, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, CPR, respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift B1.
Aerosolized Generating Procedures, B2 | At the end of shift B2, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, CPR, respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift B2.
Aerosolized Generating Procedures, B3 | At the end of shift B3, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, CPR, respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift B3.
Aerosolized Generating Procedures, B4 | At the end of shift B4, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, CPR, respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift B4.
Aerosolized Generating Procedures, B5 | At the end of shift B5, up to 12 hours
  The number of participants who entered rooms with aerosolized generating procedures (intubations, positive pressure ventilation, CPR, respiratory/airway suctioning, nebulizer treatments, nasopharyngeal aspiration) during shift B5.
Contact with respiratory/influenza symptoms, A1 | At the end of shift A1, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift A1.
Contact with respiratory/influenza symptoms, A2 | At the end of shift A2, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift A2.
Contact with respiratory/influenza symptoms, A3 | At the end of shift A3, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift A3.
Contact with respiratory/influenza symptoms, A4 | At the end of shift A4, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift A4.
Contact with respiratory/influenza symptoms, A5 | At the end of shift A5, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift A5.
Contact with respiratory/influenza symptoms, B1 | At the end of shift B1, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift B1.
Contact with respiratory/influenza symptoms, B2 | At the end of shift B2, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift B2.
Contact with respiratory/influenza symptoms, B3 | At the end of shift B3, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift B3.
Contact with respiratory/influenza symptoms, B4 | At the end of shift B4, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift B4.
Contact with respiratory/influenza symptoms, B5 | At the end of shift B5, up to 12 hours
  The number of participants who were in contact with patients with respiratory symptoms, or influenza like symptoms, while wearing the N95 mask during shift B5.
Number of patients with respiratory/influenza symptoms, A1 | At the end of shift A1, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift A1.
Number of patients with respiratory/influenza symptoms, A2 | At the end of shift A2, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift A2.
Number of patients with respiratory/influenza symptoms, A3 | At the end of shift A3, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift A3.
Number of patients with respiratory/influenza symptoms, A4 | At the end of shift A4, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift A4.
Number of patients with respiratory/influenza symptoms, A5 | At the end of shift A5, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift A5.
Number of patients with respiratory/influenza symptoms, B1 | At the end of shift B1, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift B1.
Number of patients with respiratory/influenza symptoms, B2 | At the end of shift B2, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift B2.
Number of patients with respiratory/influenza symptoms, B3 | At the end of shift B3, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift B3.
Number of patients with respiratory/influenza symptoms, B4 | At the end of shift B4, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift B4.
Number of patients with respiratory/influenza symptoms, B5 | At the end of shift B5, up to 12 hours
  The number of patients with respiratory symptoms or influenza like symptoms that a participant saw while wearing the N95 mask during shift B5.
Estimated duration with patients with respiratory/influenza symptoms, A1 | At the end of shift A1, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift A1.
Estimated duration with patients with respiratory/influenza symptoms, A2 | At the end of shift A2, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift A2.
Estimated duration with patients with respiratory/influenza symptoms, A3 | At the end of shift A3, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift A3.
Estimated duration with patients with respiratory/influenza symptoms, A4 | At the end of shift A4, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift A4.
Estimated duration with patients with respiratory/influenza symptoms, A5 | At the end of shift A5, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift A5.
Estimated duration with patients with respiratory/influenza symptoms, B1 | At the end of shift B1, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift B1.
Estimated duration with patients with respiratory/influenza symptoms, B2 | At the end of shift B2, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift B2.
Estimated duration with patients with respiratory/influenza symptoms, B3 | At the end of shift B3, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift B3.
Estimated duration with patients with respiratory/influenza symptoms, B4 | At the end of shift B4, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift B4.
Estimated duration with patients with respiratory/influenza symptoms, B5 | At the end of shift B5, up to 12 hours
  The total estimated duration in minutes of contact between a participant and patients with respiratory symptoms or influenza like symptoms during shift B5.
Distance between patients with respiratory/influenza symptoms, A1 | At the end of shift A1, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift A1. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
Distance between patients with respiratory/influenza symptoms, A2 | At the end of shift A2, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift A2. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
Distance between patients with respiratory/influenza symptoms, A3 | At the end of shift A3, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift A3. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
Distance between patients with respiratory/influenza symptoms, A4 | At the end of shift A4, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift A4. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
Distance between patients with respiratory/influenza symptoms, A5 | At the end of shift A5, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift A5. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
Distance between patients with respiratory/influenza symptoms, B1 | At the end of shift B1, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift B1. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
Distance between patients with respiratory/influenza symptoms, B2 | At the end of shift B2, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift B2. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
Distance between patients with respiratory/influenza symptoms, B3 | At the end of shift B3, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift B3. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
Distance between patients with respiratory/influenza symptoms, B4 | At the end of shift B4, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift B4. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
Distance between patients with respiratory/influenza symptoms, B5 | At the end of shift B5, up to 12 hours
  The minimum estimated distance between a participant and a patient with respiratory symptoms or influenza like symptoms during shift B5. Scaled variable in order of increasing risk: more than 6ft, less than 6ft, direct contact.
COVID-19, A1 | At the end of shift A1, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift A1.
COVID-19, A2 | At the end of shift A2, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift A2.
COVID-19, A3 | At the end of shift A3, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift A3.
COVID-19, A4 | At the end of shift A4, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift A4.
COVID-19, A5 | At the end of shift A5, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift A5.
COVID-19, B1 | At the end of shift B1, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift B1.
COVID-19, B2 | At the end of shift B2, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift B2.
COVID-19, B3 | At the end of shift B3, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift B3.
COVID-19, B4 | At the end of shift B4, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift B4.
COVID-19, B5 | At the end of shift B5, up to 12 hours
  The number of participants who were in contact with patients with confirmed COVID-19 during shift B5.
Number of COVID-19 patients, A1 | At the end of shift A1, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift A1.
Number of COVID-19 patients, A2 | At the end of shift A2, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift A2.
Number of COVID-19 patients, A3 | At the end of shift A3, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift A3.
Number of COVID-19 patients, A4 | At the end of shift A4, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift A4.
Number of COVID-19 patients, A5 | At the end of shift A5, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift A5.
Number of COVID-19 patients, B1 | At the end of shift B1, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift B1.
Number of COVID-19 patients, B2 | At the end of shift B2, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift B2.
Number of COVID-19 patients, B3 | At the end of shift B3, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift B3.
Number of COVID-19 patients, B4 | At the end of shift B4, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift B4.
Number of COVID-19 patients, B5 | At the end of shift B5, up to 12 hours
  The number of patients with confirmed COVID-19 that a participant saw during shift B5.
Completed all 5 study visits (N95 A) | At the end of shift A5, up to 60 hours
  Number of N95 A masks that completed all 5 study visits.
Completed all 5 study visits (N95 B) | At the end of shift B5, up to 60 hours
  Number of N95 B masks that completed all 5 study visits.
Failed before 5 study visits (N95 A) | At the end of shift A1-A5, up to 60 hours
  Number of N95 A masks that failed before 5 study visits.
Failed before 5 study visits (N95 B) | At the end of shift B1-B5, up to 60 hours
  Number of N95 B masks that failed before 5 study visits.
Competing event (N95 A) | Between shifts A1-A5, up to 60 hours
  Number of N95 A masks which could not be fit tested due to a competing event (lost, soiled, damaged, etc).
Competing event (N95 B) | Between shifts B1-B5, up to 60 hours
  Number of N95 B masks which could not be fit tested due to a competing event (lost, soiled, damaged, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Raven, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual participant data.